CLINICAL TRIAL: NCT06283732
Title: A Clinical Study to Assess the Effect of a Supplement on Digestive Health, Overall Well-being, and Participant Experience.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amway Corp (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20392
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Digestive System Disease
Keywords: Dietary Supplements; Digestive Health; Well-being; Energy Levels
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Supplement: Greens powder (Experimental): Participants are to consume one scoop (8.5 g) of the greens powder mixed in 8-10 oz of water every morning before breakfast for two weeks.
  Interventions: Dietary Supplement: Greens powder

INTERVENTIONS:
Dietary Supplement: Greens powder — Participants are to consume one scoop (8.5 g) of the greens powder mixed in 8-10 oz of water every morning before breakfast for two weeks.

SUMMARY:
The study aims to evaluate the effectiveness of a dietary supplement (greens powder), on improving digestive health, quality of life, energy levels, and satiety over a 14-day period. Participants, aged 18-65 and experiencing mild digestive issues, will consume the greens powder daily and report outcomes through diaries and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 18-65 years.
* Willing to comply with study requirements.
* No known allergies to the ingredients listed in the product.
* Self-reported mild digestive issues (e.g., occasional bloating, stomach discomfort, occasional constipation, or occasional diarrhea).
* Generally healthy - do not live with any uncontrolled chronic disease .

Exclusion Criteria:

* Pre-existing chronic conditions that would prevent adherence to the protocol, including oncological and psychiatric disorders.
* Known severe allergic reactions that require an Epi-Pen.
* Women who are pregnant, breastfeeding, or attempting to conceive.
* History of severe diagnosed digestive disorders (e.g., IBS, IBD, Crohn's disease) or gastrointestinal-tract surgeries.
* Unwillingness to follow the study protocol.
* Invasive medical procedure within the last three weeks or planning one during the study period.
* History of substance abuse.
* Current participation or planning to participate in another research study.
* Regular consumption of probiotics, fiber, or prebiotic supplements within 3 weeks of the study.
* Regular intake of medications that may interfere with the study or study product (e.g., anticoagulants, laxatives, sedatives, beta-blockers, anti-acids) .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Digestive Health Improvement | 14 days from the start of intervention
  Measure the change in digestive health using daily diaries and the Bristol Stool Scale (BSS).

SECONDARY OUTCOMES:
Quality of Life and Well-being Enhancement | 14 days from the start of intervention
  Assess improvements in participants' quality of life, energy levels, satiety, and overall well-being through validated questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided